CLINICAL TRIAL: NCT07287787
Title: Comparative Study of Per-oral Endoscopic Myotomy (POEM) in Treatment - naïve Achalasia Patients Versus Patients With Previous Pneumatic Dilation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Omar Zein Elabedeen Ahmed, Assistant lecturer at internal medicine department - faculty of medicine - Assiut university, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 04-2025-100435
Record Dates: First submitted 2025-11-24; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Achalasia, Esophageal
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Intervention Model Description: randomized control trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (Naïve group): Patients undergoing POEM as primary therapy. (Active Comparator)
  Interventions: Procedure: per-oral endoscopic myotomy (POEM)
- - Group II (Prior Pneumatic Dilation group):Patients undergoing POEM after failed pneumatic dilation (Active Comparator)
  Interventions: Procedure: per-oral endoscopic myotomy (POEM)

INTERVENTIONS:
Procedure: per-oral endoscopic myotomy (POEM) — Briefly, the procedure included submucosal injection at the 5-6-o'clock position entry point, and mucosal incision at the posterior wall about 8-10 cm above the esophageal-gastric junction (EGJ), entry into the tunnel by clearing submucosal fibers, and then myotomy initiating about 2 cm down from the mucosal incision and extending 2-4 cm into the cardia. Afterwards, the mucosal incision will be closed using endoclips. In special circumstances, when fibrosis or adhesions present because of prior PD, the myotomy will be located in an area of normal (fibrosis-free) tissue, and a long myotomy will be made.

SUMMARY:
The aim of this study is to compare the clinical efficacy, safety, and technical outcomes of per-oral endoscopid myotomy( POEM )in treatment-naïve achalasia patients versus patients with previous pneumatic dilation.

* Study subjects:

  1. Inclusion criteria: Adult patients diagnosed with achalasia (Chicago classification types I-III by High resolution manometry (HRM) ).
  2. Exclusion criteria:

     1. Children below 18 yr.
     2. Prior surgical myotomy.
     3. pregnancy

        Groups:
* Group I (Naïve group): Patients undergoing POEM as primary therapy.
* Group II (Prior Pneumatic Dilation group): Patients undergoing POEM after failed or relapsed pneumatic dilation.

Data analyzed included the following:

* Baseline: basic demographic information, Eckardt score , manometry(HRM) , timed barium esophagogram and history of pneumatic dilation .
* Perioperative parameters (Disease duration, Surgical time, Length of hospital stay, mucosal edema, and mucosal injuries).
* Intraoperative (mucosal perforation ,bleeding in submucosal space ,pneumoperitoneum ,pneumomediastinum,pneumothorax or incompelet myotomy )and postoperative complications (Infections,esophageal leak ,subcutaneous emphysema, GERD,esophagitis ) .
* Post procedure symptoms evaluation (Eckardt score) at 1, 3&6 months after the procedure .

Eckardt score :

It is a 12-point score which is as following :

0 1 2 3 Recent weight loss (kg) none <5 kg 5-10 kg >10 kg Dysphagia none occasional daily each meal Retrosternal chest pain none occasional daily each meal Regurgitation none occasional daily each meal

A score of ≥3 is suggestive of active achalasia.

POEM technique :

Briefly, the procedure included submucosal injection at the 5-6-o'clock position entry point, and mucosal incision at the posterior wall about 8-10 cm above the esophageal-gastric junction (EGJ), entry into the tunnel by clearing submucosal fibers, and then myotomy initiating about 2 cm down from the mucosal incision and extending 2-4 cm into the cardia. Afterwards, the mucosal incision will be closed using endoclips. In special circumstances, when fibrosis or adhesions present because of prior PD, the myotomy will be located in an area of normal (fibrosis-free) tissue, and a long myotomy will be made.

Technical success was defined as a successful completion of the entire POEM procedure. Clinical success was defined as a post-POEM Eckardt score of 3.

* Research outcome measures:

  1. Primary (main):

     Clinical success at 3 and 6 months (Eckardt score ≤ 3 )
  2. Secondary (subsidiary):
* Technical success
* Procedure time
* Intra- and post-operative complications.

Data management and analysis :

Data will be collected first in sheets, and then will be in Master sheet. Data of every patient will be coded. This will be done using SPSS. Categorical data were presented as number and percentage. Continuous data is presented as mean and standard deviation (SD) if normally distributed or median and interquartile range (IQR) if non normal distributed. Other test will be used according to the results and relations needed to be studied.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with achalasia (Chicago classification types I-III by High resolution manometry (HRM) ).

Exclusion Criteria:

* Children below 18 yr.
* Prior surgical myotomy.
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-04-15 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success at 3 and 6 months (Eckardt score ≤ 3 ) | 6 months

SECONDARY OUTCOMES:
- Technical success | 1 day ( the day of the procedure )
  the procedure will be done completely or need to do premature myotomy or to be aborted due to fibrosis or any technical problem
procedure time | 1 day ( the day of the procedure)
  compare the procedure time between the 2 groups
Intraoperative & post operative complications | up to 6 months after the procedure
  define intraoperative complications ( pneumoperitoneum, pneumothorax , mucosal perforation or bleeding ) and post operative complications ( Infections,esophageal leak ,subcutaneous emphysema, GERD,esophagitis ) and compare these complications between the 2 gruops.

IPD SHARING:
Plan to Share IPD: Undecided